CLINICAL TRIAL: NCT04908943
Title: RENEW Scleroderma: A Peer-Mentored, Web Intervention for Resilience-based, Energy Management to Enhance Wellbeing and Fatigue
Acronym: RENEW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Rheumatology Research Foundation (Other)
Responsible Party: Principal Investigator, Susan Murphy, Professor of Physical Medicine and Rehabilitation and Research, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HUM00195121
Record Dates: First submitted 2021-05-26; First posted 2021-06-01 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Scleroderma
Keywords: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Diffuse; Scleroderma, Systemic

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants and study team member who randomizes participants are blinded to participant responses at randomization. However, following assignment the blind is broken.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resilience-based, Energy Management to Enhance Wellbeing and Fatigue (RENEW) (Experimental): RENEW was created by researchers, doctors, and patients with scleroderma. It is a web-based peer-led program to help manage energy and symptoms in people who have scleroderma.
  Interventions: Behavioral: RENEW
- Waitlist (No Intervention): Participants will be asked about changes in health status, and use of any new treatments or services at 6 and 12 weeks.

INTERVENTIONS:
Behavioral: RENEW — RENEW is a 12-week, peer-led, web-based program to help people with scleroderma learn skills that can be used to manage disease symptoms and improve well-being.
  Arms: Resilience-based, Energy Management to Enhance Wellbeing and Fatigue (RENEW)

SUMMARY:
The researchers seek to understand if the Resilience-based, Energy Management to Enhance Wellbeing and Fatigue (RENEW) program helps with scleroderma symptom management and disease burden. The researchers think that those participants who receive the intervention will have clinically meaningful changes of symptom management and disease burden.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of Systemic Sclerosis (SSc), any subtype
* Report a mean score of at least 4 on the Fatigue Severity Scale; potential mean range 1-9
* Have access to a computer and an internet connection
* Are able to speak and read English.

Exclusion Criteria:

* Currently undergoing structured rehabilitation or psychological treatment.
* Other issues that preclude meaningful participation in study procedures (e.g. concurrent or complex medical issues, inability to access RENEW intervention, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2021-08-28 (Actual); Primary Completion 2023-05-29 (Actual); Study Completion 2023-05-29 (Actual)

PRIMARY OUTCOMES:
Change in Fatigue | Up to 12 weeks
  Fatigue is measured by The Functional Assessment of Chronic Illness Therapy (FACIT) -Fatigue 13a. FACIT is a questionnaire with 13 questions and a score ranging from 13-65. Higher scores indicate greater fatigue.

SECONDARY OUTCOMES:
Change in Pain Interference | Up to 12 weeks
  Pain interference is measured by Patient-Reported Outcomes Measurement Information System (PROMIS) pain interference 4a scale Pain Interference 4a will assess self-reported consequences of pain with 4 questions ranked on a 5-point scale, from "not at all" to "very much". The minimum score is 4 and the maximum score is 20. Lower scores suggest less pain interference.
Change in Resilience | Up to 12 weeks
  Resilience is measured by Connor-Davidson Resilience Scale 10 (CD-RISC-10). It is a 10 item self-report rating scale 0 (not true at all) to 4 (true nearly all the time). The overall score range from 0 (no resilience) to 40 (High Resilience).
Change in Depressive symptoms | Up to 12 weeks
  Depressive symptoms are measured by PROMIS depression 4a assesses self-reported negative mood (e.g., sadness), views of self (e.g., worthlessness), social cognition (e.g., loneliness), and decreased positive affect and engagement. Items are all answered on a 5-point scale from 1=Never to 5=Always. Scores can range from 0 meaning no anxiety/depression to 40 meaning high

CONTACTS AND LOCATIONS:
Overall Officials: Susan Murphy, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified data that underlie the results reported in the article will be shared with researchers who present a methodologically sound proposal.
Supporting Information: Study Protocol
Time Frame: Data will be available beginning 9 months and ending 36 month after publication of primary analyses.
Access Criteria: Proposals should be directed to sumurphy@med.umich.edu. To gain access, data requesters will need to sign a data use agreement at which time the researchers will provide access to the dataset. After 36 months, data will be deposited at the Inter-university Consortium for Political and Social Research (ICPSR) at the University of Michigan
URL: http://www.icpsr.umich.edu/

REFERENCES:
- [Derived] Chen YT, Hassett AL, Khanna D, Murphy SL. Resilience partially mediates the association between perceived social isolation and life satisfaction in people with systemic sclerosis. J Scleroderma Relat Disord. 2024 Jun;9(2):154-161. doi: 10.1177/23971983241232853. Epub 2024 Mar 5. PMID 38910596
- [Derived] Chen YT, Hassett AL, Huang S, Khanna D, Murphy SL. Peer-Led Symptom Management Intervention to Enhance Resilience in People With Systemic Sclerosis: Mediation Analysis From a Randomized Clinical Trial. Arthritis Care Res (Hoboken). 2024 Sep;76(9):1278-1286. doi: 10.1002/acr.25352. Epub 2024 May 31. PMID 38622109
- [Derived] Chen YT, Harper AE, Phanhdone T, Alore M, Hicks S, Pape A, Jay GM, Bolde S, Feldpausch J, Guetterman TC, Khanna D, Murphy SL. Impact of a resilience-building energy management intervention for people with systemic sclerosis: a mixed methods study. Rheumatol Adv Pract. 2024 Mar 8;8(2):rkae040. doi: 10.1093/rap/rkae040. eCollection 2024. PMID 38618141
- [Derived] Murphy SL, Chen YT, Alore M, Hicks S, Pape A, Hassett AL, Kratz AL, Whibley D, Harper AE, Huang S, Jay G, Bolde S, Khanna D. Effects of a Resilience-Building Energy Management Program on Fatigue and Other Symptoms in Systemic Sclerosis: A Randomized Controlled Trial. Arthritis Care Res (Hoboken). 2024 Mar;76(3):318-327. doi: 10.1002/acr.25253. Epub 2024 Jan 12. PMID 37846437